CLINICAL TRIAL: NCT03477214
Title: Tactile Imaging and Electromyography of Female Pelvic Floor
Brief Title: Tactile Imaging and Electromyography
Status: Completed | Type: Observational
Sponsor: Advanced Tactile Imaging, Inc. (Industry)
Collaborators: Princeton Urogynecology (Other)
Responsible Party: Sponsor
Other Study IDs: TIEMG08
Record Dates: First submitted 2018-02-15; First posted 2018-03-26 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Urinary Incontinence; Overactive Bladder
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Normal: No UI, no OAB conditions. Transvaginal biomechanical and electromyography mapping will be completed.
  Interventions: Diagnostic Test: Biomechanical and electromyography mapping
- Urinary incontinence: Urinary incontinence conditions. Transvaginal biomechanical and electromyography mapping will be completed.
  Interventions: Diagnostic Test: Biomechanical and electromyography mapping
- Overactive bladder: Overactive bladder conditions
  Interventions: Diagnostic Test: Biomechanical and electromyography mapping

INTERVENTIONS:
Diagnostic Test: Biomechanical and electromyography mapping — The vaginal tactile imaging probe will acquire biomechanical and electromyography high definition measurements for anterior and posterior compartments along entire vagina.

SUMMARY:
Urinary incontinence (UI) and overactive bladder (OAB) in women has high prevalence which is increasing with the age. In adults aged 40 and older in the US demonstrated prevalence rate of 27.2% among man and 43.1% among women, respectively. Urine Incontinence was reported to affect 15% of women ages 40 to 49, 25% ages 60 to 69, and 38% of women age 80 and older.

DETAILED DESCRIPTION:
Pelvic floor disorders result from neuro-urinary pathology as well as muscle functional impairment due to changes in bio-mechanical properties of soft tissues with the age. That is why pelvic floor characterization and diagnosis must include electomyographic (EMG) and biomechanical measurements (pressure) or better if EMG and tactile imaging with improved spatial resolution. The quantitative and objective imaging data for pelvic floor conditions could allow an effective treatment of OAB and UI.

In this research the investigators propose to develop a new device for accurate diagnosis of the diseased conditions by measuring the pelvic floor muscles strength and EMG activity. The value to society is high given by the prevalence of OAB and UI.

ELIGIBILITY:
Inclusion Criteria:

* Women above age of 21 with normal pelvic floor condition for the control
* Women with SUI conditions as defined by International Continence Society guidelines
* Women with OAB conditions as defined by American Urological Association and Society of Urodinamics, Female Pelvic Medicine & Urogenital Reconstruction.

Exclusion Criteria:

* Any prior pelvic floor surgery related to SUI, POP or OAB conditions
* Active skin infection or ulceration within the vagina
* Presence of the vaginal septum
* Active cancer of the colon, rectum wall, cervix, vaginal, uterus or bladder
* Ongoing radiation therapy for pelvic cancer; impacted stool
* Surgically absent rectum or bladder
* Sever hemorrhoids
* Significant circulatory or cardiac conditions that could cause excessive risk
* Significant pre-existing pelvic pain including levator ani syndrome, severe vaginismus or vulvodynia.

Min Age: 21 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: There is no inclusion or exclusion criteria based on ethnic background, religion, or other division of population other than these stated in Exclusion Criteria section.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-12-24 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Transvaginal biomechanical maps | Four months
  Transvaginal biomechanical maps (pressures in Pa) will be recorded and compared for UI and OAB versus normal conditions.
Transvaginal electromyography maps | Four months
  Transvaginal electromyography maps (electrical voltages in mV) will be recorded and compared for UI and OAB versus normal conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Heather van Raalte, MD, Study Director — Princeton Urogynecology
Locations (2):
- United States (2):
  - Princeton Urogynecology, Princeton, New Jersey
  - Institute of Female Pelvic Medicine & Reconstructive Surgery (IFPM), Allentown, Pennsylvania